CLINICAL TRIAL: NCT01376232
Title: Open Label Study to Assess the Pharmacokinetics of GSK1278863A Coadministered With a High Fat Meal or an Inhibitor of CYP2C8 (Gemfibrozil)
Brief Title: Study to Assess the Pharmacokinetics of GSK1278863A Coadministered With a High Fat Meal or an Inhibitor of CYP2C8 (Gemfibrozil)
Acronym: DDI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Octagon Research Solutions, Incoporated (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 113634
Record Dates: First submitted 2011-06-16; First posted 2011-06-20 (Estimated); Last update posted 2017-06-09 (Actual); Status verified 2017-06

CONDITIONS: Anaemia
Keywords: Anaemia; Drug- Drug Interaction
MeSH Terms: conditions — Anemia | interventions — GSK1278863; Food; Gemfibrozil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- GSK1278863 (Experimental): 100 mg of GSK1278863
  Interventions: Drug: GSK1278863
- GSK1278863 + food (Experimental): 100 mg of GSK1278863 given with a high fat meal
  Interventions: Drug: GSK1278863 + food
- GSK1278863 + Gemfibrozil (Experimental): GSK1278863A 100mg + Gemfibrozil 600mg steady state
  Interventions: Drug: Gemfibrozil

INTERVENTIONS:
Drug: GSK1278863 — GSk1278863 100mg
  Arms: GSK1278863
Drug: GSK1278863 + food — High Fat meal + 100 mg GSK1278863
  Arms: GSK1278863 + food
Drug: Gemfibrozil — 600 mg Gemfibrozil
  Arms: GSK1278863 + Gemfibrozil

SUMMARY:
Study to Assess the Pharmacokinetics of GSK1278863A Coadministered with a High Fat Meal or an Inhibitor of CYP2C8 (gemfibrozil),]

DETAILED DESCRIPTION:
The purpose of this study is to assess the clinical drug-drug interaction potential of GSK1278863A with medications that are inhibitors of CYP2C8 enzyme in order to support co-administration of similar agents in later phase development. Specifically. this study will assess the pharmacokinetics of a single dose of GSK1278863A administered alone or co-administered with gemfibrozil, a potent inhibitor of CYP2C8, following steady-state oral administration of gemfibrozil. Finally, to support the co-administration of GSK1278863A with food, this study will assess the pharmacokinetics of a single oral dose of GSK1278863A under fasting conditions and following a standard high-calorie, high fat meal.

ELIGIBILITY:
Inclusion Criteria:

* AST, ALT, alkaline phosphatase and bilirubin > 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%)
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures
* Male or female between 18 and 55 years of age inclusive, at the time of signing the informed consent
* A female subject is eligible to participate if she is of:Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol < 40 pg/ml (<140 pmol/L) is confirmatory]. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods in Section 8.1 if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2-4 weeks should elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method
* Male subjects must agree to use one of the contraception methods listed in Section 8.1. This criterion must be followed from the time of the first dose of study medication until 5 terminal half-lives post-last dose
* Body weight < 50 kg and BMI within the range 19 - 29.9 kg/m2 (inclusive)
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form
* QTcB or QTcF < 450 msec; or QTc < 480 msec in subjects with Bundle Branch Block

Exclusion Criteria:

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* The values of hematological parameters at screening are: Any values outside the reference range
* A positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines
* The values of the following tests at screening are: Serum ferritin: outside the reference range
* A positive test for HIV antibody
* Clinically significant CPK >3 X ULN or deemed clinically significant by the investigator
* Calculated creatinine clearance: < 80 mL/min
* Subjects with a pre-exisisting condition interfering with normal gastrointestinal anatomy or motility, and/or hepatic function-that could interfere with the absorption, metabolism, and/or excretion of the study drugs. Examples of conditions that could interfere with normal gastriointestinal anatomy or motility include cholecystectomy, vagotomy, malabsorption, Crohn's disease, ulcerative colitis, or celiac sprue
* History of regular alcohol consumption within 6 months of the study defined as: an average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 g of alcohol: a half-pint (~240 ml) of beer, 1 glass (125 ml) of wine or 1 (25 ml) measure of spirits
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 12 weeks, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer)
* History of peptic ulcer disease
* History of malignancy tumor. Non-melanoma skin cancer that has been definitely removed is allowed
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 14 days or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period
* Pregnant females as determined by positive serum or urine hCG test at screening or prior to dosing
* Lactating females
* Unwillingness or inability to follow the procedures outlined in the protocol
* Subject is mentally or legally incapacitated
* History of sensitivity to heparin or heparin-induced thrombocytopenia
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening
* Consumption of red wine, apples, star fruit, or citrus fruits/juices including blood oranges (with the exception of oranges, mandarins and lemons) from 7 days prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor this will not interfere with the study procedures and compromise subject safety

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2010-11-08 (Actual); Primary Completion 2010-12-20 (Actual); Study Completion 2010-12-20 (Actual)

PRIMARY OUTCOMES:
GSK1278863A (and metabolites, as appropriate) AUC(0-¥) and Cmax | 48 hours
  1. To assess the relative bioavailability GSK1278863A following single-dose administration under fasting and fed (standard high fat/calorie meal) conditions

SECONDARY OUTCOMES:
1. Plasma GSK1278863A (and metabolites, as appropriate) AUC(0-t), tmax, and t1/2. | 48hr
  1. To assess the safety and tolerability of GSK1278863A when coadministered with a high-fat meal and steady-state gemfribrozil
Adverse event, clinical laboratory, ECG, vital signs, and concurrent medication assessments. | 48 hours and duration of study
  Safety and tolerability parameters

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Electronics City, Bengalore, India

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 113634 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/113634?search=study&search_terms=113634#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 113634 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113634 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113634 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113634 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113634 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113634 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113634 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register